CLINICAL TRIAL: NCT04643431
Title: Risk Assessment of Carotid Plaques Based on Pressure Estimation Using 3D Contrast-enhanced Ultrasound
Brief Title: Risk Assessment of Carotid Plaques Using 3D Contrast-Enhanced Ultrasound
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB #20D.699
Record Dates: First submitted 2020-11-19; First posted 2020-11-25 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2024-07

CONDITIONS: Carotid Atherosclerosis
MeSH Terms: conditions — Carotid Artery Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Carotid SHAPE estimation (Experimental): The ultrasound contrast agent is infused (4-10 mL/min). An area within the plaque demonstrating internal flow is selected and a software based calibration algorithm is executed. After selecting the optimal acoustic output power 3D SHAPE volumes of the entire plaque (including the carotid artery) are acquired. Infusion is stopped and after microbubble clearance a second set of 3D SHAPE volumes (without contrast) are obtained.
  Interventions: Diagnostic Test: Perflutren

INTERVENTIONS:
Diagnostic Test: Perflutren — The ultrasound contrast agent is used to improve the quality of ultrasound imaging and is infused over 5-10 minutes. The contrast agent consists of the gas-filled microbubbles smaller than the capillary size which circulate in the vascular system. The contrast agent is cleared from the body naturally within 30 minutes.
  Other Names: SHAPE with Definity

SUMMARY:
This is an open-label, non-randomized study conducted at Thomas Jefferson University comparing pressure-gradient estimates (obtained between a carotid plaque and the carotid artery) to imaging and histology markers of plaque vulnerability. There is an inverse relationship between the subharmonic signal magnitude from contrast-enhanced ultrasound microbubbles and ambient pressure. This pressure estimation technique (referred as SHAPE) will be used to estimate the pressure gradient across the carotid plaque cap noninvasively in vivo.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years old and willing and able to participate. Patients with atherosclerosis scheduled for carotid endarterectomy

Exclusion Criteria:

* • Pregnancy or breast-feeding at the time of the scan

  * Patients with known hypersensitivity or allergy to any component (including perflutren) of Definity (Lantheus Medical Imaging, Billerica, MA).
  * Patients who are medically unstable, patients who are seriously or terminally ill, and patients whose clinical course is unpredictable. For example:

    * Patients on life support or in a critical care unit.
    * Patients with unstable occlusive disease (e.g., crescendo angina).
    * Patients with clinically unstable cardiac arrhythmias, such as recurrent ventricular tachycardia.
    * Patients with uncontrolled congestive heart failure (NYHA Class IV).
    * Patients with recent cerebral hemorrhage.
    * Patients who have undergone surgery within 24 hours prior to the study sonographic examination.
  * Patients with unstable cardiopulmonary conditions (acute myocardial infarction, acute coronary artery syndromes, worsening or unstable congestive heart failure, or serious ventricular arrhythmias) or respiratory distress syndrome.
  * Patients with uncontrollable emphysema, pulmonary vasculitis, pulmonary hypertension or a history of pulmonary emboli.
  * Patients who have received any contrast medium (X-ray, MRI, CT or ultrasound) in the 24 hours prior to the research ultrasound exam

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2023-04-05 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Correlation between the pressure gradient and surrogate (imaging and histological) predictors | pre-endarterectomy
  The estimates of pressure-gradient across the plaque cap from 3D SHAPE technique will be compared with the surrogate imaging and histological predictors using Pearson's correlation coefficient. The correlations between the surrogate predictors will be also calculated using Pearson's correlation coefficient. We expect the pressure-gradient estimates from SHAPE technique is moderately correlated (above 0.5) with the surrogate predictors.

CONTACTS AND LOCATIONS:
Overall Officials: Kibo Nam, PhD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas jefferson University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No